CLINICAL TRIAL: NCT05983861
Title: Risk Factors for Multidrug Resistant Bacteria at ICU Admission
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: José Raimundo Araujo de Azevedo (Other)
Responsible Party: Sponsor-Investigator, José Raimundo Araujo de Azevedo, ICU Assistent Physician, Hospital Sao Domingos
Organization: Hospital Sao Domingos (Other)
Other Study IDs: 17/2023
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Multi Drug Resistant Bacteria
Keywords: Infection; Multi drug Resistant bacteria; Risk Factors; Critical Care; Score
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multi drug resistant group: All critically ill adult patients (with no exclusion criteria) admitted to the ICU with microbiological confirmed diagnosis of infection at admission and multi drug resistant bacteria isolation :
  Interventions: Diagnostic Test: Identification o Multi Drug Resistant Bacteria
- Multi sensible bacteria group: All critically ill adult patients (with no exclusion criteria) admitted to the ICU with microbiological confirmed diagnosis of infection at admission and multi drug sensible bacteria isolation :
  Interventions: Diagnostic Test: Identification o Multi Drug Resistant Bacteria

INTERVENTIONS:
Diagnostic Test: Identification o Multi Drug Resistant Bacteria — Identification o Multi Drug Resistant Bacteria

SUMMARY:
The objective of this single-center prospective observational study is to evaluate possible independent risk factors for multidrug-resistant (MDR) bacteria upon ICU admission by analyzing comorbidities, epidemiological data, and laboratory/microbiological information of the subjects.

DETAILED DESCRIPTION:
Background: Infection is one of the main reason for a patient to be admitted to an intensive care unit (ICU) and it's fundamental to use the right antibiotic as soon as possible, possibly needing broad-spectrum antibiotics. However, the main problem is that widening the spectrum of drugs will generate pressure on the hospital microbiota, leading to the development of multi-drug resistant bacteria

Purpose: A large number of ICU-admitted patients have infection/sepsis as their major problem, requiring treatment with antibiotics. With knowledge of the presumed risk factors for antibiotic resistance, the assistant physician could use broad-spectrum drugs with greater certainty.

Objectives: Our objective will be to evaluate risk factors for infection caused by multi-drug resistant germs upon ICU admission and assess the severity of the disease in comparison to patients infected with susceptible bacteria. Ultimately, we aim to develop and validate a clinical tool to assist physicians in selecting the appropriate antibiotic for their patients

Methods: An observational prospective study with a control group will be conducted, including all patients admitted to the ICU with an infectious disease initiated within 48 hours of hospital admission and with a positive microbiologic result. Patients with isolation of only susceptible bacteria will be allocated to the control group, while patients with MDR bacteria will be assigned to the study group, referred to as the MDR group. The data to be collected will include sex, age, previous use of antibiotics in the last three months, previous hospital admissions, previous isolation of MDR germs, sensitivity profile of the isolated germs, severity of disease (measured by SAPS 3), presence of sepsis diagnosis at admission, length of stay in the ICU, and 28-day mortality

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the ICU with an infectious disease initiated within 48 hours of hospital admission and a microbiological positive result for bacteria

Exclusion Criteria:

* Patients with results considered as contamination according to the institutional protocol.
* Surgical wound and bloodstream infections.
* Microbiological isolation of only fungi.
* Vigilance cultures, such as anal, rectal, nasal, and axillary swabs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICU with an infectious disease initiated within 48 hours of hospital admission and with a positive microbiologic result.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Determine risk factors for multi-drug resistant germs in ICU admission. | 28 days
  Analysis of resistance profile of germs and patient's comorbidities to determine the risk factors for drug resistance.

SECONDARY OUTCOMES:
Mortality between control and case group | 28 days
  Compare mortality in 28 days between patients with infection caused by MDR bacteria and non-resistant bacteria.
Mean LOS of each group | 28 days
  Compare the length of stay in ICU between the control and case groups.
Severity between groups using SAPS 3 | 28 days
  Compare the severity of disease between groups using the SAPS 3 score.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niederman MS, Baron RM, Bouadma L, Calandra T, Daneman N, DeWaele J, Kollef MH, Lipman J, Nair GB. Initial antimicrobial management of sepsis. Crit Care. 2021 Aug 26;25(1):307. doi: 10.1186/s13054-021-03736-w. PMID 34446092
- [Result] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781
- [Result] Bassetti M, Rello J, Blasi F, Goossens H, Sotgiu G, Tavoschi L, Zasowski EJ, Arber MR, McCool R, Patterson JV, Longshaw CM, Lopes S, Manissero D, Nguyen ST, Tone K, Aliberti S. Systematic review of the impact of appropriate versus inappropriate initial antibiotic therapy on outcomes of patients with severe bacterial infections. Int J Antimicrob Agents. 2020 Dec;56(6):106184. doi: 10.1016/j.ijantimicag.2020.106184. Epub 2020 Oct 9. PMID 33045353
- [Result] Kalil AC, Johnson DW, Lisco SJ, Sun J. Early Goal-Directed Therapy for Sepsis: A Novel Solution for Discordant Survival Outcomes in Clinical Trials. Crit Care Med. 2017 Apr;45(4):607-614. doi: 10.1097/CCM.0000000000002235. PMID 28067711
- [Result] Liu VX, Fielding-Singh V, Greene JD, Baker JM, Iwashyna TJ, Bhattacharya J, Escobar GJ. The Timing of Early Antibiotics and Hospital Mortality in Sepsis. Am J Respir Crit Care Med. 2017 Oct 1;196(7):856-863. doi: 10.1164/rccm.201609-1848OC. PMID 28345952
- [Result] Wong D, Wong T, Romney M, Leung V. Comparative effectiveness of beta-lactam versus vancomycin empiric therapy in patients with methicillin-susceptible Staphylococcus aureus (MSSA) bacteremia. Ann Clin Microbiol Antimicrob. 2016 Apr 26;15:27. doi: 10.1186/s12941-016-0143-3. PMID 27112143
- [Result] Fernandez-Martinez NF, Carcel-Fernandez S, De la Fuente-Martos C, Ruiz-Montero R, Guzman-Herrador BR, Leon-Lopez R, Gomez FJ, Guzman-Puche J, Martinez-Martinez L, Salcedo-Leal I. Risk Factors for Multidrug-Resistant Gram-Negative Bacteria Carriage upon Admission to the Intensive Care Unit. Int J Environ Res Public Health. 2022 Jan 18;19(3):1039. doi: 10.3390/ijerph19031039. PMID 35162062